CLINICAL TRIAL: NCT01200004
Title: A Phase I Study of Epigenetic Immunomodulation Through the Use of Azacitidine, Lenalidomide, and Grifola Frondosa in Patients With Advanced Malignancy
Brief Title: Study of Grifola Frondosa (Maitake), Azacitidine, and Lenalidomide
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Yukiguni Maitake Company Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0076
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Cancers
Keywords: Advanced solid tumor; Azacitidine; Grifola frondosa; Basidiomycete fungus; Lenalidomide
MeSH Terms: interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Azacitidine + Lenalidomide (Experimental): Azacitidine 75 mg/m2 subcutaneous or by vein on days 1 - 5 of a 28 day cycle. Lenalidomide starting dose 10 mg by mouth daily on days 1-21 of a 28 day cycle, until maximum tolerated dose (MTD) reached. MTD used for combination and expansion groups.
  Interventions: Drug: Azacitidine; Drug: Lenalidomide
- Azacitidine + Lenalidomide + Grifola Frondosa (Experimental): Once Lenalidomide MTD identified in combination with azacitidine, Grifola frondosa added. Cycle 1, azacitidine on day 1, lenalidomide on day 2 and Grifola frondosa on day 3. Azacitidine daily for 5 days every 28 days while lenalidomide and Grifola frondosa on days 1-21 of subsequent cycles.
  Interventions: Drug: Azacitidine; Drug: Lenalidomide; Drug: Grifola Frondosa
- Expansion Group A (Experimental): Azacitidine + Lenalidomide MTD, then 2 weeks later Grifola frondosa
  Interventions: Drug: Lenalidomide
- Expansion Group B (Experimental): Azacitidine + Grifola Frondosa, then 2 weeks later Lenalidomide
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m2 subcutaneous or by vein on days 1 - 5 of a 28 day cycle.
  Other Names: 5-Azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Azacitidine + Lenalidomide; Azacitidine + Lenalidomide + Grifola Frondosa
Drug: Lenalidomide — Starting dose 10 mg by mouth daily on days 1-21 of a 28 day cycle, until maximum tolerated dose (MTD) reached. MTD used for combination and expansion groups.
  Other Names: CC-5013; Revlimid
Drug: Grifola Frondosa — 3 mg/kg by mouth twice a day on days 1 - 21 of a 28 day cycle.
  Arms: Azacitidine + Lenalidomide + Grifola Frondosa

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of Grifola frondosa extract, azacitidine, and lenalidomide that can be given to patients with advanced cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Azacitidine is designed to block certain proteins in cancer cells whose job is to stop the function of the tumor-fighting proteins. By blocking the "bad" proteins, the tumor-fighting genes may be able to work better.

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may decrease the growth of cancer cells.

Grifola frondosa extract is a natural substance taken from maitake mushrooms. Researchers want to learn if it can cause the body's immune system to react against cancer.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to receive either azacitidine and lenalidomide, azacitidine and Grifola frondosa, or azacitidine, lenalidomide, and Grifola frondosa at a dose level based on when you joined this study.

Up to 4 dose levels of azacitidine and lenalidomide will be tested. Up to 2 dose levels of azacitidine and Grifola frondosa will be tested. At the beginning of the study, 3-6 participants will be enrolled at each dose level of the study drug combinations. The first group of participants will receive the lowest dose level of azacitidine and lenalidomide. Each new group will receive a higher dose of the study drug combination than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found. After enrollment in the azacitidine and lenalidomide group is completed, the next group of participants will receive the lowest dose level of azacitidine and Grifola frondosa. Each new group will receive a higher dose of the study drug combination than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found.

After the highest dose of the azacitidine and lenalidomide or Grifola frondosa combinations are found, new participants enrolling in this study will begin receiving Grifola frondosa along with azacitidine and lenalidomide. Up to 2 dose levels will be tested. The first group of participants will receive the lowest dose level of lenalidomide. The next group will receive a higher dose of lenalidomide than the group before it, if no intolerable side effects were seen. The doses of azacitidine and Grifola frondosa will stay the same.

The dose of the study drug combination that you receive may be lowered if you have any intolerable side effects.

Study Drug Administration:

A study drug "cycle" is 28 days.

On Days 1-5 of each Cycle, you will receive azacitidine either under the skin or by vein. If you receive azacitidine as an injection under the skin, you will receive it over 10 minutes. If you receive azacitidine by vein, you will receive it over 40 minutes.

On Day 2 of Cycle 1, you will begin taking lenalidomide 1 time each day until Day 21, then you will have a 7 day-rest period. For Cycle 2 and every cycle after that, you will take lenalidomide 1 time each day on Days 1-21 followed by a 7-day rest period. Lenalidomide is a capsule that you will take by mouth with water. The capsules should be swallowed whole. You should not break, chew, or open the capsules.

If you are assigned to receive Grifola frondosa, you will also begin taking Grifola frondosa 2 times each day on Day 2 of Cycle 1 if you are also taking azacitidine. If you are also taking azacitidine and lenalidomide, you will begin taking Grifola frondosa on Day 3 of Cycle 1. Depending on the dose level you are assigned to, you will either take Grifola frondosa 2 times each day until Day 21 followed by a 7-day rest period, or you will take Grifola frondosa 2 times daily during all cycles. Grifola frondosa is a liquid extract that comes in a glass bottle. Your dose of Grifola frondosa will be based on when you joined the study and your body weight.

Expansion Groups:

After the highest tolerable dose of each study drug combination is found, 42 additional participants will be enrolled in 3 expansion groups (14 in each group), one group for each study drug combination at the highest tolerable dose or a dose level that has been shown to be safe.

Study Visits:

The following tests and procedures will be performed within 7 days before your first dose of study drug:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.

Women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test within 10 to 14 days before the first dose of the study drug combination and again within 24 hours before receiving lenalidomide.

Before you begin each cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* You will be asked about any side effects you may be having.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.
* Women who are able to have children will have a blood pregnancy test.

Every week during Cycles 1 and 2, blood (about 2 teaspoons) will be drawn for routine tests.

Women who are able to have children will have a blood (about 1 teaspoon) pregnancy test every week during Cycle 1.

At the end of every 2 cycles (Cycles 2, 4, 6, and so on), you will have a CT, MRI, PET scan, and/or x-ray to check the status of the disease.

If you are in the one of the Expansion Groups, blood (about 6 teaspoons each time) will be drawn for biomarker testing before you take the first dose of study drug, on Days 21 and 28 of Cycle 1, 1 time during each cycle after that, and at the end-of-study visit.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

Within 30 days after your last dose of the study drug combination, you will have an end-of-study visit. The following tests and procedures performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* You will be asked about any side effects you may be having.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.
* If the study doctor thinks it is needed, you will have a chest x-ray, CT, MRI, and/or PET scan to check the status of the disease.
* Women who are able to have children will have a blood pregnancy test.

This is an investigational study. Grifola frondosa extract is not FDA approved for any usage. Its use in this study is investigational. Azacitidine and lenalidomide are FDA approved and commercially available for the treatment of multiple myeloma and myelodysplastic syndrome. The use of the study drug combination (Grifola frondosa, azacitidine, and lenalidomide) is currently being used for research purposes only.

Up to 102 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed diagnosis of an advanced solid tumor refractory to standard treatment or for which no standard therapy is available.
2. Patients must have ECOG performance status 2 or better (0-2).
3. Patients must have normal organ and marrow function as defined: Absolute lymphocyte count > 1,000 /uL, Absolute neutrophil count > 1,500 /uL, Platelets > 75,000 /uL, Bilirubin </= 1.5 * ULN and AST and/or ALT </= 2.5 * the institutional upper limit of normal (ULN), </= 5 * ULN for patients with liver metastases, Serum creatinine within normal limits; if abnormal, then a calculated creatinine clearance >/= 50 mL/min
4. Patients must be able to understand and be willing to sign an IRB-approved written informed consent document.
5. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mlU/mL within 10-14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
6. Patients must be 18 years of age or older since the safety and dosages of these study drugs has not been demonstrated in the pediatric population. Exception: patients who are 13 years old or older and have more than 50 kg of body weight will be eligible after consultation with their pediatric attending.
7. Life expectancy greater than 3 months based on the attending physician's discretion.
8. All study participants must be registered in the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, symptomatic cardiac arrhythmia, active bleeding, active thrombosis, or psychiatric illness/social situations that would limit compliance with study requirements.
2. History of stroke or transient ischemic attack within 6 months prior to study enrollment and significant vascular disease (e.g., aortic aneurysm, aortic dissection) and symptomatic peripheral vascular disease.
3. History of allergic reactions to the study drugs or their analogs.
4. Patients that have had any treatment specific for tumor control within 3 weeks of study drug treatment or: a. within 2 weeks if cytotoxic agents were given weekly b. within 6 weeks for nitrosoureas or mitomycin C c. within 4 half-lives for targeted agents with half lives and pharmacodynamic effects lasting less than 5 days (that includes, but is not limited to, erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents) d. failed to recover from toxic effects of any therapy prior to study entry
5. Concurrent known immunosuppressors.
6. Inability to swallow oral medication.
7. Pregnant or breastfeeding women.
8. Concurrent enrollment on another research study.
9. Known hepatitis B and C infection, HIV infection and autoimmune disorders.
10. Subjects with known moderate or severe renal impairment will be excluded if creatinine clearance < 60 ml/min.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks
  MTD defined by patient dose limiting toxicities (DLTs) that occur in the first cycle (4 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org